CLINICAL TRIAL: NCT05257733
Title: Evaluation of the Diagnostic Contributions of Nerve Ultrasound in Chronic Inflammatory Demyelinating Polyneuropathy Associating Systemic Diseases
Brief Title: Evaluation of the Diagnostic Contributions of Nerve Ultrasound in Chronic Inflammatory Demyelinating Polyneuropathy Associating Systemic Diseases (CIDP Echo-nerf)
Acronym: CIDP echo-nerf
Status: Withdrawn | Type: Observational
Why Stopped: Departure of the project leader
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2022/II-01
Record Dates: First submitted 2022-02-15; First posted 2022-02-25 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CIDP associated with systemic diseases: Patients with CIDP associated with systemic diseases
  Interventions: Other: None, pure observationnal study
- CIDP without systemic diseases: Patients with CIDP without other systemic diseases
  Interventions: Other: None, pure observationnal study

INTERVENTIONS:
Other: None, pure observationnal study — pure observationnal study

SUMMARY:
Chronic inflammatory demyelinating polyradiculoneuritis (CIDP) is an autoimmune disorder of the peripheral nervous system, most commonly affecting the myelin sheath. The pathophysiology of CIDP is not completely understood, but both humoral and cellular immunity appear to be involved in the genesis of this disease. Some diseases are particularly associated with CIDP such as diabetes, monoclonal gammopathies and hematological diseases.

CIDP can occur before, after or simultaneously with the onset of systemic diseases. The systemic diseases most often seen in association with polyneuropathies are lupus, Gougerot-Sjögren's syndrome and sarcoidosis.

Ultrasound of peripheral nerves is a useful and accessible tool. In CIDP, this examination can reveal diffuse or segmental nerve hypertrophy. In addition to the size of the nerve, this exploration analyzes the echogenicity and the aspect of the different fascicles within the nerve. S. Goedee et al have shown that nerve ultrasound has very good diagnostic parameters and low interobserver variability in the diagnosis of CIDP. F. Härtig et al suggests that nerve ultrasound can predict the therapeutic response and describes 3 main patterns: hypoechoic enlargement (active inflammation), nerve enlargement with hyperechoic add-on fascicles (axonal degeneration) and almost no enlargement ("cured" CIDP).

DETAILED DESCRIPTION:
CIDP may be progressive or relapsing, most frequently clinically symmetric, sensorimotor with proximal and distal involvement developing over at least 8 weeks but variants as distal, multifocal, focal, motor or sensory CIDP have been also described. Cell-mediated and humoral mechanisms act together in an aberrant immune response to cause damage to peripheral nerves but, by molecular mimicry it causes other autoimmune system diseases. This paper focuses on the intersection of CIDP and other autoimmune disease with an emphasis on shared pathology and mutually characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed at Nîmes University Hospital between 2012 and 2021
* Age > 18 years
* Diagnosis of definite CIDP or possible CIDP according to the new EFNS/PNS 2021 criteria
* Diagnosis of definite CIDP/CIDP possible with systemic diseases and respectively diagnosis of definite CIDP/CIDP possible for the control group confirmed by electroneuromyography, concordant with the clinical examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed at Nîmes University Hospital between 2012 and 2021 with CIDP
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Median nerve cross-sectional area | Base line, Day 0
  Comparison of median nerve cross-sectional area on nerve ultrasound in patients with definite PIDC/PIDC with associated systemic disease with that of patients with PIDC/PIDC without systemic disease
ulnar nerve at wrist cross-sectional area | Base line, Day 0
  Comparison of ulnar nerve at wrist cross-sectional area on nerve ultrasound in patients with definite PIDC/PIDC with associated systemic disease with that of patients with PIDC/PIDC without systemic disease
ulnar at mid-arm nerve cross-sectional area | Base line, Day 0
  Comparison of ulnar nerve at mid-arm cross-sectional area on nerve ultrasound in patients with definite PIDC/PIDC with associated systemic disease with that of patients with PIDC/PIDC without systemic disease
ulnar nerve at elbow cross-sectional area | Base line, Day 0
  Comparison of ulnar nerve at elbow cross-sectional area on nerve ultrasound in patients with definite PIDC/PIDC with associated systemic disease with that of patients with PIDC/PIDC without systemic disease
radial nerve cross-sectional area | Day of diagnosis of CIDP
  Comparison of radial nerve cross-sectional area on nerve ultrasound in patients with definite PIDC/PIDC with associated systemic disease with that of patients with PIDC/PIDC without systemic disease
superficial radial branch nerve cross-sectional area | Base line, Day 0
  Comparison of superficial radial branch nerve cross-sectional area on nerve ultrasound in patients with definite PIDC/PIDC with associated systemic disease with that of patients with PIDC/PIDC without systemic disease
vagus nerve cross-sectional area | Base line, Day 0
  Comparison of vagus nerve cross-sectional area on nerve ultrasound in patients with definite PIDC/PIDC with associated systemic disease with that of patients with PIDC/PIDC without systemic disease
C6 root nerve cross-sectional area | Base line, Day 0
  Comparison of C6 root nerve cross-sectional area on nerve ultrasound in patients with definite PIDC/PIDC with associated systemic disease with that of patients with PIDC/PIDC without systemic disease
C5 root nerve cross-sectional area | Base line, Day 0
  Comparison of C5 root nerve cross-sectional area on nerve ultrasound in patients with definite PIDC/PIDC with associated systemic disease with that of patients with PIDC/PIDC without systemic disease
sural nerve cross-sectional area | Base line, Day 0
  Comparison of sural nerve cross-sectional area on nerve ultrasound in patients with definite PIDC/PIDC with associated systemic disease with that of patients with PIDC/PIDC without systemic disease
superficial fibula nerve cross-sectional area | Base line, Day 0
  Comparison of superficial fibula nerve cross-sectional area on nerve ultrasound in patients with definite PIDC/PIDC with associated systemic disease with that of patients with PIDC/PIDC without systemic disease
tibial nerve at ankle cross-sectional area | Base line, Day 0
  Comparison of tibial nerve at ankle cross-sectional area on nerve ultrasound in patients with definite PIDC/PIDC with associated systemic disease with that of patients with PIDC/PIDC without systemic disease
popliteal nerve cross-sectional area | Base line, Day 0
  Comparison of popliteal nerve cross-sectional area on nerve ultrasound in patients with definite PIDC/PIDC with associated systemic disease with that of patients with PIDC/PIDC without systemic disease
fibular nerve at neck cross-sectional area | Base line, Day 0
  Comparison of fibular nerve at neck cross-sectional area on nerve ultrasound in patients with definite PIDC/PIDC with associated systemic disease with that of patients with PIDC/PIDC without systemic disease
fibular at supra-neck nerve cross-sectional area | Base line, Day 0
  Comparison of fibular at supra-neck nerve cross-sectional area on nerve ultrasound in patients with definite PIDC/PIDC with associated systemic disease with that of patients with PIDC/PIDC without systemic disease

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, France

REFERENCES:
- [Result] Schmidt B, Toyka KV, Kiefer R, Full J, Hartung HP, Pollard J. Inflammatory infiltrates in sural nerve biopsies in Guillain-Barre syndrome and chronic inflammatory demyelinating neuropathy. Muscle Nerve. 1996 Apr;19(4):474-87. doi: 10.1002/(SICI)1097-4598(199604)19:43.0.CO;2-9. PMID 8622727
- [Result] Sommer C, Koch S, Lammens M, Gabreels-Festen A, Stoll G, Toyka KV. Macrophage clustering as a diagnostic marker in sural nerve biopsies of patients with CIDP. Neurology. 2005 Dec 27;65(12):1924-9. doi: 10.1212/01.wnl.0000188879.19900.b7. PMID 16380614
- [Result] Spies JM, Westland KW, Bonner JG, Pollard JD. Intraneural activated T cells cause focal breakdown of the blood-nerve barrier. Brain. 1995 Aug;118 ( Pt 4):857-68. doi: 10.1093/brain/118.4.857. PMID 7655884
- [Result] Madia F, Frisullo G, Nociti V, Conte A, Luigetti M, Del Grande A, Patanella AK, Iorio R, Tonali PA, Batocchi AP, Sabatelli M. pSTAT1, pSTAT3, and T-bet as markers of disease activity in chronic inflammatory demyelinating polyradiculoneuropathy. J Peripher Nerv Syst. 2009 Jun;14(2):107-17. doi: 10.1111/j.1529-8027.2009.00220.x. PMID 19691533
- [Result] Press R, Pashenkov M, Jin JP, Link H. Aberrated levels of cerebrospinal fluid chemokines in Guillain-Barre syndrome and chronic inflammatory demyelinating polyradiculoneuropathy. J Clin Immunol. 2003 Jul;23(4):259-67. doi: 10.1023/a:1024532715775. PMID 12959218
- [Result] Mei FJ, Ishizu T, Murai H, Osoegawa M, Minohara M, Zhang KN, Kira J. Th1 shift in CIDP versus Th2 shift in vasculitic neuropathy in CSF. J Neurol Sci. 2005 Jan 15;228(1):75-85. doi: 10.1016/j.jns.2004.10.001. Epub 2004 Nov 12. PMID 15607214
- [Result] Kurihara M, Kurata Y, Sugimoto I, Hatanaka Y, Sakurai Y. High PR3-ANCA positivity in a patient with chronic inflammatory demyelinating polyneuropathy. eNeurologicalSci. 2016 Oct 5;6:4-5. doi: 10.1016/j.ensci.2016.10.001. eCollection 2017 Mar. PMID 29260006
- [Result] Greenberg SA. P-ANCA vasculitic neuropathy with 12-year latency between onset of neuropathy and systemic symptoms. BMC Neurol. 2002 Oct 31;2(1):10. doi: 10.1186/1471-2377-2-10. PMID 12437775
- [Result] Abraham H, Kuzhively J, Rizvi SW. Chronic Inflammatory Demyelinating Polyneuropathy (CIDP): An Uncommon Manifestation of Systemic Lupus Erythematosus (SLE). Am J Case Rep. 2017 Sep 12;18:980-983. doi: 10.12659/ajcr.903541. PMID 28894082
- [Result] Siddiqui K, Cahalane E, Keogan M, Hardiman O. Chronic ataxic neuropathy with cold agglutinins: atypical phenotype and response to anti-CD20 antibodies. Neurology. 2003 Nov 11;61(9):1307-8. doi: 10.1212/wnl.61.9.1307. No abstract available. PMID 14610153
- [Result] Rodriguez Y, Vatti N, Ramirez-Santana C, Chang C, Mancera-Paez O, Gershwin ME, Anaya JM. Chronic inflammatory demyelinating polyneuropathy as an autoimmune disease. J Autoimmun. 2019 Aug;102:8-37. doi: 10.1016/j.jaut.2019.04.021. Epub 2019 May 6. PMID 31072742
- [Result] Wolbert J, Cheng MI, Meyer zu Horste G, Su MA. Deciphering immune mechanisms in chronic inflammatory demyelinating polyneuropathies. JCI Insight. 2020 Feb 13;5(3):e132411. doi: 10.1172/jci.insight.132411. PMID 32051341
- [Result] Seeliger T, Prenzler NK, Gingele S, Seeliger B, Korner S, Thiele T, Bonig L, Suhs KW, Witte T, Stangel M, Skripuletz T. Neuro-Sjogren: Peripheral Neuropathy With Limb Weakness in Sjogren's Syndrome. Front Immunol. 2019 Jul 11;10:1600. doi: 10.3389/fimmu.2019.01600. eCollection 2019. PMID 31354737